CLINICAL TRIAL: NCT00250393
Title: Placebo-Controlled , Crossover , Double-Blind Study of KW-6002(Istradefylline) in the Treatment of Parkinson's Disease. [Monotherapy]
Brief Title: A Study of Istradefylline (KW-6002) for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-0407
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; monotherapy
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
To establish the efficacy of 40 mg/day doses of istradefylline for the change in Unified Parkinson's Disease Rating Scale (UPDRS) part-III (Motor examination) score in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
To establish the efficacy of 40mg/d doses of istradefylline for the change in UPDRS part-III (Motor examination) score in patients with Parkinson's disease (PD). Patients who meet entry criteria will be randomly assigned to receive study drug in 1 of 2 arms: Condition A (doses of 40mg/d istradefylline) in Period 1 followed by Condition B (matching placebo) in Period 2 (putting 4 weeks interval phase between two periods ) or Condition B in Period 1 followed by Condition A in Period 2(putting 4 weeks interval phase between two periods ). Patients will be participated for 12 weeks and will have interim visits and end of treatment visit to assess the efficacy and safety of istradefylline.

ELIGIBILITY:
Inclusion Criteria:

1. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD.
2. PD stages 1-3 for Modified Hoehn and Yahr Scale.
3. Be at least 30 years of age.

Exclusion Criteria:

1. Neurosurgical treatment for PD.
2. History of psychosis.
3. Diagnosis of cancer within 5 years.
4. Diagnosis of clinically significant illness of any organ system.
5. Mini-mental status examination score of 25 or less.
6. Taking any excluded medications.
7. History of drug or alcohol abuse or dependence within the past two years.
8. History of seizures or neurological malignant syndrome.
9. Clinical depression.
10. Pregnant or lactating females.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of 40mg/d doses of istradefylline for the change in UPDRS part-III (Motor examination) score in patients with Parkinson's disease (PD).

SECONDARY OUTCOMES:
To evaluate the efficacy of 40mg/d dose of istradefylline for the change in UPDRS part-I (Mentation, behavior and mood), part-II (Activities of daily living) score and UPDRS total (parts I-III) score.
To evaluate change in the Clinical Global Impression - Improvement scale (CGI-I).
To evaluate change in the Clinical Global Impression - Severity of Illness scale (CGI-S).
To evaluate the safety of 40mg/d doses of istradefylline.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan